CLINICAL TRIAL: NCT00033280
Title: A Phase II Trial Of Pre-Irradiation And Concurrent Temozolomide In Patients With Newly Diagnosed Anaplastic Oligodendrogliomas And Mixed Anaplastic Oligoastrocytomas
Brief Title: Temozolomide Plus Radiation Therapy in Treating Patients With Newly Diagnosed Anaplastic Oligodendrogliomas or Mixed Anaplastic Oligoastrocytomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-BR-0131; CDR0000069270
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2018-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic oligodendroglioma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Glioma | interventions — Temozolomide; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pre-RT temozolomide, RT plus temozolomide (Experimental): Pre-radiation therapy (RT) temozolomide, RT plus temozolomide
  Interventions: Drug: temozolomide; Procedure: neoadjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: temozolomide
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining temozolomide with radiation therapy in treating patients who have newly diagnosed anaplastic oligodendrogliomas or mixed anaplastic oligoastrocytomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the rate of progression in patients with newly diagnosed anaplastic oligodendrogliomas or mixed anaplastic oligoastrocytomas treated with neoadjuvant and concurrent temozolomide with radiotherapy.
* Determine the toxicity of this regimen in these patients.
* Determine the survival of patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to response to neoadjuvant temozolomide (stable disease or partial response (PR) vs complete response (CR)).

Patients receive oral temozolomide on days 1-7 and 15-21. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with CR or PR receive 2 courses beyond CR or PR.

Within 6 weeks after completion of neoadjuvant temozolomide, patients with stable disease or PR undergo radiotherapy 5 days a week for 6.5 weeks. Patients also receive oral temozolomide daily for 42 days concurrently with radiotherapy.

Patients with CR after completion of neoadjuvant temozolomide undergo observation.

Patients are followed at 9 and 12 months, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 37 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed supratentorial pure or mixed anaplastic oligodendroglioma

  * Unifocal or multifocal disease
  * Prior suspected or proven low-grade glioma eligible provided biopsy reveals pure or mixed anaplastic oligodendroglioma that has not been previously treated with radiotherapy and/or chemotherapy
* No equivocal oligodendroglial element
* No tumors predominantly located in the posterior fossa (i.e., brainstem or cerebellum)
* No spinal cord tumors
* No evidence of spinal drop metastasis or spread to noncontiguous meninges

PATIENT CHARACTERISTICS:

Age:

* 18 to 65

Performance status:

* Zubrod 0-1

Life expectancy:

* More than 12 weeks

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 2 times normal
* Aspartate aminotransferase (AST) no greater than 3 times normal
* Alkaline phosphatase no greater than 2 times normal

Renal:

* Creatinine no greater than 1.5 times normal

Other:

* No active infection
* No other medical problems that would preclude study participation
* No other malignancy within the past 3 years except carcinoma in situ of the cervix or nonmelanoma skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior chemotherapy for this malignancy
* No prior temozolomide

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to the brain, head, or neck

Surgery:

* At least 14 days since prior surgery requiring general anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2002-07; Primary Completion 2005-04 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Rate of progression at 6 months (post-chemotherapy/pre-irradiation progression) | From start of treatment to 6 months

SECONDARY OUTCOMES:
Overall Survival | From registration to date of death or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Vogelbaum, MD, PhD, Study Chair — The Cleveland Clinic
Locations (39):
- United States (38):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - Monmouth Medical Center, Long Branch, New Jersey
  - Wayne Memorial Hospital, Inc., Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Anderson Area Cancer Center, Anderson, South Carolina
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Saint John Regional Hospital, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vogelbaum MA, Berkey B, Peereboom D, Macdonald D, Giannini C, Suh JH, Jenkins R, Herman J, Brown P, Blumenthal DT, Biggs C, Schultz C, Mehta M. Phase II trial of preirradiation and concurrent temozolomide in patients with newly diagnosed anaplastic oligodendrogliomas and mixed anaplastic oligoastrocytomas: RTOG BR0131. Neuro Oncol. 2009 Apr;11(2):167-75. doi: 10.1215/15228517-2008-073. Epub 2008 Sep 8. PMID 18779504
- [Result] Vogelbaum MA, Berkey B, Peereboom D, et al.: RTOG 0131: phase II trial of pre-irradiation and concurrent temozolomide in patients with newly diagnosed anaplastic oligodendrogliomas and mixed anaplastic oligodendrogliomas: relationship between 1p/19q status and progression-free survival. [Abstract] J Clin Oncol 24 (Suppl 18): A-1517, 2006.
- [Result] Vogelbaum MA, Berkey B, Peereboom D, et al.: RTOG 0131: phase II trial of pre-irradiation and concurrent temozolomide in patients with newly diagnosed anaplastic oligodendrogliomas and mixed anaplastic oligodendrogliomas. [Abstract] J Clin Oncol 23 (Suppl 16): A-1520, 119s, 2005.